CLINICAL TRIAL: NCT02848989
Title: Qigong Mind-Body Exercise For Persistent Post-Surgical Pain In Breast Cancer Survivors: A Pilot Study
Brief Title: Qigong For PPSP In Breast Cancer Pain In Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Dr., M.D., Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-347
Record Dates: First submitted 2016-06-01; First posted 2016-07-29 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer Surgery Pain; Breast Cancer; Stage 0-III Breast Cancer
Keywords: Breast Cancer Surgery Pain; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qigong Mind-Body Exercise (QMBE) (Experimental): After the screening procedures confirm that you are eligible to participate in the research study:
  * Breast cancer survivors with persistent post-surgical pain (PPSP) into a 12-week program of Qigong mind-body exercise (QMBE).
  * Outcome assessments related to pain, function, and quality of life
  Interventions: Other: Qigong Mind-Body Exercise

INTERVENTIONS:
Other: Qigong Mind-Body Exercise — An exercise program that involves gentle movements combined with breathing/relaxation techniques

SUMMARY:
Studies have shown that on-going pain following breast surgery is common and may limit the ability to participate in physical activity, cause tiredness, difficulty in daily chores/activities as well as other problems.

This study is evaluating whether participating in a 12-week Qigong program (pronounced chee kung), an exercise program that involves gentle movements combined with breathing/relaxation techniques, also known as mind-body exercise, leads to improvement of pain, physical function, and quality of life among breast cancer survivors that have significant pain following surgery.

DETAILED DESCRIPTION:
This is a pilot/feasibility study designed to look at the potential benefits of a 12-week program of Qigong mind-body exercise program. The study applies to women who have completed physical therapy treatment on symptoms such as pain, and difficulty moving/strength of arm in women who are experiencing on-going symptoms after breast cancer surgery. The results of this study will be used to help design future studies of the effect of Qigong programs in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage 0-III breast cancer;
* Persistent post-surgical pain at least 3 months after completion of surgery, chemotherapy, and/or radiation;
* Completion of a course of physical therapy

Exclusion Criteria:

* Unstable cardiovascular disease in the last 6 months
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g. untreated major depression or psychosis, substance abuse, severe personality disorder);
* Metastatic breast or other cancer;
* Participation in more than 240 minutes of moderate-intensity exercise per week (as determined by Leisure Score Index questionnaire)
* Pregnant or breastfeeding
* Recent history of attending regular QMBE or similar classes (e.g. yoga or tai chi classes), (i.e.20 or more classes in the past 6 months).
* Currently enrolled in a physical therapy course

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Rate of completion of QMBE intervention | 12 months
  Complete recruitment of target enrollment of 21 participants within 12 month timeframe.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
  Total number of adverse events sustained from participation in QMBE will be collected for each participant through home practice logs for at home QMBE participation and instructors will report any adverse events that occur during QMBE class on attendance logs. Any adverse events observed will be evaluated according to the DFCI/Harvard Cancer Center guidelines. The study will be considered safe if zero adverse events are observed/reported from participation in prescribed QMBE classes and/or at home practice.

SECONDARY OUTCOMES:
Changes in Quality of life | 6 months
  QOL will be assessed using the Functional Assessment of Cancer Therapy Breast Symptom Index (FACT-B+4). This instrument consists of 42 items that measure physical, emotional, social and functional well-being, as well as breast cancer specific symptomology associated with upper extremity dysfunction.
Degree of Pain | 6 months
  Degree of pain will be measured by the Brief Pain Inventory Short Form (BPI SF) and a Pain Medication Log.21 The BPI SF consists of 9 items that measure the severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. Reliability coefficients for the BPI Severity and Interference scales ranged from .82 to .95
Grip Strength | 3 months
  Grip strength of both hands will be assessed using the Jamar® Hand Dynamometer. Measurement will be recorded to the nearest 0.5 kg, and repeated an average of three times
Gait & Postural Control | 3 months
  Gait & postural control will be kinematically assessed during standing and walking using an 8-camera motion analysis system (Vicon 512, Oxford, UK) using standard protocols employed in prior mind-body studies as well as clinical evaluations for both children and adults with walking abnormalities due to mobility-limiting conditions, at the Motion Analysis Laboratory at Spaulding Rehabilitation Hospital.
Pain Catastrophizing | 3 months
  Pain catastrophizing scale will be used to assess catastrophic thinking associated with pain. This instrument consists of 13 items that measure rumination, magnification, and helplessness related to pain.
Shoulder Strength | 3 months
  Will be assessed using manual muscle testing (MMT).
Range of Motion | 3 months
  Will be assessed using standard goniometric measurement.
Fatigue | 3 months
  Fatigue will be assessed by the 13 item FACIT-F fatigue subscale. This validated instrument measures the intensity of fatigue experienced during the 7 days before questionnaire administration.
Self-esteem | 3 months
  Self-esteem will be measured by the 10 item Rosenberg Self-Esteem Scale. This validated instrument measures global self-worth by measuring both positive and negative feelings about the self.
Anxiety & Depression | 3 months
  Anxiety and depression will be measured by the Hospital and Anxiety and Depression Scale (HADS). This validated instrument consists of 14 items that measure current feelings of anxiety and depression.
Stress Levels | 3 months
  Stress levels will be measured by the 10 item Perceived Stress Scale (PSS). This validated instrument measures the degree to which situations in one's life are appraised as stressful.
Mindfulness | 3 months
  Mindfulness will be assessed using the Multidimensional Assessment of Interoceptive Awareness Scale (MAIA). This 32-item instrument measures a patient's bodily and emotional awareness and ability to self-regulate these factors.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No